CLINICAL TRIAL: NCT06029881
Title: Validation of a New Non-intrusive Technology for Detecting Sleep Apnea
Brief Title: Portable System for Non-intrusive Monitoring of Sleep
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erasme University Hospital (Other)
Collaborators: Fonds de la Recherche Scientifique (fnrs) (Unknown)
Responsible Party: Principal Investigator, Philippe Van de Borne, Professor, Erasme University Hospital
Other Study IDs: B4062023000020
Record Dates: First submitted 2023-08-16; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Sleep Apnea
Keywords: obstructive sleep apnea; Ballistocardiography; Seismocardiography; Polysomnography; sleep assessment
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obstructive sleep apnea patients: Patients admitted for complaints of sleep disturbances with no prior significant cardiovascular disease.
  Inclusion criteria:
  * 18 < age <70
  * BMI < 35 kg/m2
  Exclusion criteria:
  * Being under any kind of OSA treatment (cPAP therapy, etc.)
  * Having been diagnosed with Atrial fibrillation, significant valvular heart disease, or ventricular dysfunction
  * Age <18 or age > 70
  * BMI > 35 kg/m2
  Interventions: Device: Movesense MD

INTERVENTIONS:
Device: Movesense MD — This device can be attached to the skin (on the chest and center of mass) during sleep using a belt and adhesive electrodes.

SUMMARY:
Obstructive sleep apnea (OSA) is a prevalent kind of sleep-disordered breathing affecting one-seventh of the world's population. Almost 45 percent of this population suffers from mild to severe apnea. However, in many cases it remains undiagnosed, leading to increased health risks. Sleep-disordered breathing, as seen in OSA, can have serious long-term consequences, including sympathetic nervous system activation, sleep disturbances, heart remodeling, and cardiovascular disease development.

Polysomnography is the standard method for assessing sleep-breathing disorders, which requires the attachment of various sensors by a trained technician or a healthcare professional. However, if the diagnosis of OSA depends on referral to a sleep laboratory, and if the referral is reliant on symptoms of an OSA syndrome, then current screening approaches may exclude a large population of individuals at risk. Besides, the number of sleep centers and caregivers is limited, and the associated costs are high. Therefore, alternative techniques allowing home monitoring are necessary.

The goal of this observational study is to evaluate the accuracy of the Kinocardiography technique in detecting apneic episodes during sleep and comparing the results with the gold standard polysomnography in 47 patients suffering from obstructive sleep apnea. We hypothesize that this device is able to detect sleep-disordered breathing events, and thus to compute the apnea-hypopnea index, with an accuracy that is close to that of the polysomnography.

Participants who meet the criteria will be invited to participate in this protocol and do both polysomnography and kinocardiography records simultaneously at night during sleep.

DETAILED DESCRIPTION:
1. Study Glossary

   * BCG = Ballistocardiography
   * ECG = Electrocardiography
   * PSG = Polysomnography
   * SCG = Seismocardiography
   * KCG = Kinocardiography
2. Monitoring Technique

   Ballistocardiography (BCG) and seismocardiography (SCG) are two promising technologies for monitoring vital signs during sleep. BCG measures body movements caused by blood flow ejection at each cardiac contraction, while SCG detects micro-vibrations from heart contractions on the chest surface. These low-cost and unobtrusive technologies have been used in various sleep studies, showing promise in vital sign recording, detecting abnormal breathing episodes, and studying the effects of disease and environmental conditions. However, more research and replication of studies are required for widespread application.

   Kinocardiography:

   Kinocardiography (KCG) is a technique that combines BCG and SCG with electrocardiography (ECG). The BCG module is placed close to the subject's center of mass in the lumbar vertebrae. The SCG module is placed on the sternum beneath the clavicle, close to the heart and major blood vessels. Each module is a MOVESENSE device that incorporates a three-axis accelerometer and three-axis gyroscope sensor and is attached to the body using standard sticky gel electrodes and a belt. The overall system is remotely controlled via a Bluetooth-connected smartphone or tablet. This device allows the measurement of the micro-accelerations induced by the cardiac activity at the body's surface. By computing these accelerations, it is possible to calculate other parameters, such as the kinetic energies associated with the contraction of the heart.

   Polysomnography:

   Polysomnography (PSG) includes various techniques to monitor neurophysiological, cardiopulmonary, and other physiologic parameters simultaneously. PSG uses electroencephalogram, electrooculogram, electromyogram, ECG, pulse oximetry, airflow, and respiratory effort to identify the underlying causes of sleep disturbances.
3. Safety Reporting

   The MOVESENSE device will be used in this study to collect ECG and signals from accelerometers and gyroscopes. Once this data has been collected, then the analysis will be conducted within the Erasme hospital. This device is a CE-marked medical device (https://ec.europa.eu/tools/eudamed/#/screen/search-device/8d619c90-794a-4564-9a54-829aefa9c707).

   The hazard probability is extremely low, and its severity is minimal (the only possibility is feeling uncomfortable with the electrodes' gel on the skin).

   If a subject becomes uncomfortable, they can call the nurse/operator throughout the measurement and will be able to let the operator know right away if they want to stop the measurement.
4. Strategies for participant recruitment

The recruitment will be done among the subjects referred for PSG as required by their medical condition. This study will not affect in any manner the regular medical care of the patients admitted to the sleep laboratory. Subjects will be recruited within the routine of the sleep laboratory in the Erasme hospital. Subjects who meet the criteria will be invited to participate in this protocol and do both PSG and KCG records simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* The participants should be adult patients who come to Erasme Hospital's sleep department with complaints about sleep disturbances.
* 18 < age <70
* BMI < 35 kg/m2

Exclusion Criteria:

* Being under any kind of obstructive sleep apnea treatment (cPAP therapy, etc.)
* Having been diagnosed with Atrial fibrillation, significant valvular heart disease, or ventricular dysfunction
* Age <18 or age > 70
* BMI > 35 kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for complaints of sleep disturbances with no prior treatment for sleep apnea and no known cardiovascular pathologies.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of MOVESENSE sensor in detecting patients suffering from apnea | During 1 night (~8hours)
  Sensitivity and Specificity of MOVESENSE sensor in detecting patients suffering from apnea based on the apnea-hypopnea index (AHI) and different grades of severity: AHI<5; 5<AHI<15; 15<AHI<30; 30<AHI.

SECONDARY OUTCOMES:
Variation of kinetic energy during apneic episodes | During 1 night (~8hours)
  Measurement of changes in seismocardiography/ballistocardiography integral of kinetic energy (in mJ.s) during and immediately after an apneic episode.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe van de Borne, Principal Investigator — Professor
Locations (1):
- Erasme hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No